CLINICAL TRIAL: NCT06488261
Title: A Long-Term Follow-Up Safety Study of Subjects With Gaucher Disease Who Previously Received AVR-RD-02
Brief Title: Long Term Follow-Up for Safety of AVR-RD-02
Status: Active, not recruiting | Type: Observational
Sponsor: John Bernat (Other)
Responsible Party: Sponsor-Investigator, John Bernat, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202309221
Record Dates: First submitted 2023-11-20; First posted 2024-07-05 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects who received AVR-RD-02: Subjects who received AVR-RD-02 in a separate parent trial
  Interventions: Biological: AVR-RD-02

INTERVENTIONS:
Biological: AVR-RD-02 — No study drug is administered in this study. Subjects who received AVR-RD-02 in a separate parent trial will be evaluated in this trial for long-term safety.

SUMMARY:
The goal of this observational study is to assess the safety and tolerability of AVR-RD-02 treatment in subjects who previously received AVR-RD-02 treatment (single dose administration).

DETAILED DESCRIPTION:
Subjects who received AVR-RD-02 in the preceding treatment study (NCT04145037) and who meet all eligibility criteria may participate. Subjects will be asked to return for study visits annually for 14 years to assess measures of safety and persistence of AVR-RD-02 treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria for participation in this study:

1. Subject must be willing and able to provide written informed consent for the JAB-GD-001 study in accordance with applicable regulations and guidelines and to comply with all study visits and procedures.
2. Subject must have been enrolled in the preceding AVROBIO AVRO-RD-02-201 treatment study and have received AVR-RD-02 treatment

Exclusion Criteria

Subject has any medical, psychological, or other condition that, in the opinion of the Investigator:

* Might interfere with the subject's participation in the study (including consenting to procedures); and/or
* Poses any additional risk to the subject; and/or
* Might confound the results of any study-required assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Gaucher disease who previously received the investigational gene therapy product AVR-RD-02
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2037-06 (Estimated); Study Completion 2037-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of newly diagnosed malignancy, hematologic disorder, and/or autoimmune or rheumatologic disorder | Baseline to Year 14
Change from baseline over time in hemoglobin concentration | Baseline to Year 14
Change from baseline over time in platelet count | Baseline to Year 14

SECONDARY OUTCOMES:
Change from baseline over time in glucocerebrosidase (GCase) enzyme activity in whole blood | Baseline to Year 14
Average vector copy number (VCN) from whole blood using quantitative polymerase chain reaction (qPCR) analysis | Baseline to Year 14
Change from baseline over time in anti-GCase total antibodies and subsequent titers | Baseline to Year 14
Identification of potential aberrant clonal expansion(s) assessed by performing insertional site analysis (ISA) from whole blood | Baseline to Year 14
Presence of replication competent lentivirus (RCL) | Baseline to Year 14

CONTACTS AND LOCATIONS:
Overall Officials: John A. Bernat, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States